CLINICAL TRIAL: NCT01490216
Title: Open-Label Pilot Study of Lisdexamfetamine for Treatment of Cocaine Dependence
Brief Title: Pilot Study of Lisdexamfetamine for Treatment of Cocaine Dependence
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3002-11961-00006857
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Cocaine Dependence
Keywords: cocaine; lisdexamfetamine; vyvanse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lisdexamfetamine (Other): open label
  Interventions: Drug: lisdexamfetamine

INTERVENTIONS:
Drug: lisdexamfetamine — 20mg q.d. to 70mg b.i.d
  Other Names: vyvanse

SUMMARY:
The purpose of this study is to evaluate ideal dose or lisdexamfetamine and tolerability, plus reduction in cocaine use and craving.

DETAILED DESCRIPTION:
Evaluate ideal dose or lisdexamfetamine and tolerability, plus reduction in cocaine use and craving as determined by self-report and cocaine-positive urine samples.

ELIGIBILITY:
.Inclusion Criteria:

1. Men and women between the ages of 18-65 who meet Diagnostic and Statistical Manual -IV criteria for current cocaine dependence
2. Used cocaine at least four days in the past month
3. Individuals must be in good general health
4. Individuals must be capable of giving informed consent and capable of complying with study procedures
5. Women of child-bearing age must agree to use a method of contraception with proven efficacy, consisting of one of the following: 1) Any form of hormonal contraception; 2) Intra-uterine device; 3) Sterilization; 4) Double-barrier contraception which is a combination of two of the following: condoms, spermicide, diaphragm. Pregnancy tests will be performed monthly and if a woman becomes pregnant, the study medication will be discontinued.

Exclusion Criteria:

1. Individuals who meet DSM-IV-TR criteria for bipolar disorder, schizophrenia, or any psychotic disorder other than transient psychosis due to drug abuse
2. Individuals with any other current Axis I psychiatric disorder as defined by DSM-IV-TR that in the investigator's judgment are unstable, or would be disrupted by study medication, or are likely to require pharmacotherapy during the study period
3. Individuals physiologically dependent on any other drugs (excluding nicotine or cannabis) which require medical intervention
4. Individuals with current psychostimulant abuse or dependence (other than cocaine dependence)
5. Individuals with current suicidal risk
6. Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms
7. Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension (SBP > 140, diastolic blood pressure > 90, or heart rate > 100 when sitting quietly), acute hepatitis (patients with chronic mildly elevated transaminases (< 3x upper limit of normal are acceptable), or uncontrolled diabetes
8. Individuals with a history of seizures, hyperthyroidism and/or glaucoma
9. History of allergic reaction to study medication
10. Women who are pregnant or nursing
11. Currently being prescribed psychotropic medication by another physician (other than sleep medication)
12. Individuals who are legally mandated (e.g., to avoid incarceration) to participate in substance abuse treatment program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
maximum total lisdexamfetamine dose achieved during the study period defined as the highest amount of medication per day maintained for a seven day period | Study weeks 3-6

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Mooney, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States